CLINICAL TRIAL: NCT02000609
Title: Phase II, Partial Blind, Randomized, Placebo Controlled, 5-way Cross-over Study to Evaluate the Pharmacodynamics of BDP(Beclomethasone Diproprionate)/B17MP (Beclomethasone-17-Monoproprionate) and FORMOTEROL FUMARATE (FF) Across Two Different Dose Levels of CHF 1535 NEXThaler DPI (Dry Powder Inhaler) and CHF 1535 pMDI (Pressurized Metered-dose Inhaler)in Adult COPD (Chronic Obstructive Pumonary Disease) Patients
Brief Title: A Phase II, 5-way Cross-over Study to Evaluate the Pharmacodynamics of "Nexthaler" Dry Powder Inhaler in COPD Patients
Acronym: NEXThaler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-01535BC1-02
Record Dates: First submitted 2013-11-21; First posted 2013-12-04 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: COPD
Keywords: pharmacodynamics COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- CHF 1535 NEXThaler 800/48 ug (Active Comparator): single dose administration of CHF 1535 100/6 NEXThaler DPI, total dose: 800ug BDP, 48 ug Formoterol Fumarate
  Interventions: Drug: CHF 1535 NEXThaler 800/48
- CHF 1535 NEXThaler PLACEBO (Placebo Comparator): single dose administration of placebo via NEXThaler DPI
  Interventions: Drug: CHF 1535 NEXThaler PLACEBO
- CHF 1535 pMDI 200/12 (Active Comparator): single dose administration of CHF 1535 100/6 pMDI , total dose: 200 ug BDP, 12 ug Formoterol Fumarate
  Interventions: Drug: CHF 1535 pMDI 200/12
- CHF 1535 100/6 pMDI 800/48 (Active Comparator): single dose administration of CHF 1535 100/6 pMDI total dose: 800ug BDP, 48 ug Formoterol Fumarate
  Interventions: Drug: CHF1535 pMDI 800/48
- CHF 1535 NEXThaler 200/12 (Active Comparator): single dose administration of CHF 1535 100/6 pMDI, total dose: 200 ug BDP, 12 ug Formoterol Fumarate
  Interventions: Drug: CHF 1535 NEXThaler 200/12

INTERVENTIONS:
Drug: CHF 1535 NEXThaler 800/48
  Arms: CHF 1535 NEXThaler 800/48 ug
Drug: CHF 1535 NEXThaler 200/12
  Arms: CHF 1535 NEXThaler 200/12
Drug: CHF 1535 NEXThaler PLACEBO
  Arms: CHF 1535 NEXThaler PLACEBO
Drug: CHF 1535 pMDI 200/12
  Arms: CHF 1535 pMDI 200/12
Drug: CHF1535 pMDI 800/48
  Arms: CHF 1535 100/6 pMDI 800/48

SUMMARY:
The study aim is to compare the pharmacodynamic effects (cardiovascular effects- primary variable: Heart rate over 4 hours post dosing- ) after administration of BDP and formoterol administered as CHF 1535 100/6 NEXThaler DPI or CHF1535 pMDI at two different dose levels.

DETAILED DESCRIPTION:
The effects of both formulations on serum potassium and serum glucose and the general safety and tolerability of study treatments will be also evaluated

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (≥ 40 and ≤ 75 years old).
* Outpatients with diagnosis of moderate/severe stable COPD, according to GOLD (Global Initiative for Chronic Obstructive Lung Disease) guidelines update 2013 at least in the 6 months before the screening visit.
* A post-bronchodilator FEV1(Forced Expiratory Volume in one second) ≥ 40 and < 80% of the predicted normal value and FEV1/FVC (Forced Vital Capacity) < 0.7, after 4 puffs (4 x 100 µg) of salbutamol pMDI. If this criterion is not met at screening, the test can be repeated once before commencing of the run-in period.
* Ability to use pMDI (pressured metered-dose inhaler)and DPI (dry powder Inhaler) devices
* Current or past smoker of at least 10 pack/years where one pack-year is equivalent to 20 cigarettes per day for 1 year

Exclusion Criteria:

* Pregnant or lactating female subjects.
* Current diagnosis of Asthma (as defined by the current GINA (Global Initiative for Asthma guidelines 2012 (update), or history of allergic rhinitis.
* COPD exacerbations requiring systemic steroids and /or antibiotics and/or oral or nebulized beta 2-agonists in the 4 weeks prior to screening and until randomization.
* Lower Respiratory Tract Infection (LRTI) in the 4 weeks prior to screening and until randomization.
* Patients with serum potassium levels < 3.5 mEq/L (milliequivalent per liter).
* History of substance abuse or drug abuse within 12 months prior to screening visit.
* Known respiratory disorders other than COPD including but not limited to α1 antitrypsin deficiency, active tuberculosis, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, restrictive lung disease and interstitial lung disease.
* Intolerance or contra-indication to treatment with beta 2-agonists and/or inhaled corticosteroids or allergy to any component of the study treatments.
* Patients treated with non-cardioselective β-blockers in the month preceding the screening visit or during the study period.
* Patients who have clinically significant cardiovascular disease according to investigator's judgement. Thus includes but is not limited to:

  * congestive heart failure (NYHA class > 3);
  * acute ischemic heart disease within the past 12 months of screening;
  * Sustained cardiac arrhythmias (supraventricular or ventricular, >30 seconds duration) at or within 6 months of screening;
  * Non sustained cardiac arrhythmias (supraventricular or ventricular, > 3 beats < 30 seconds and or ending spontaneously and or asymptomatic);
  * History of sustained and non-sustained cardiac arrhythmias (supraventricular or ventricular);
  * 2nd or 3rd degree Atrioventricular conduction block;
  * Left Bundle Branch Block.
* An abnormal 12-lead ECG (QRS> 120 msec, PR> 220 msec, HR < 40 bpm, Heart Rate > 110 bpm) at screening or at randomization.
* Patients whose electrocardiogram (12-lead ECG) shows QTcF >450 ms for males or QTcF > 470 ms for females at screening or at randomisation.
* Patients whose DBP/SBP is higher than: DBP 90 mmHg or SBP 160 mmHg at screening or at randomization.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Average 4-hour Heart Rate bpm (beats per minutes) | 4 hours

SECONDARY OUTCOMES:
QTcF (QT interval Fridericia's formula corrected) (milliseconds), QRS (milliseconds) and PR (milliseconds) intervals, PAC (Premature Atrial Contraction- percentage) burden, PVC (Premature Ventricular Contraction-percentage) burden, Blood Pressure (mmHg) | -45, -30, -15min pre-dose, 5, 10, 20, 30, 45min, 1, 1.5, 2, 3, 4, 5, 5, 7, 8, 10 12 hr post dose

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Principal Investigator — Medicine Evaluation Unit, Manchester (UK)
Locations (1):
- Medicine Evaluation Unit, Manchester, United Kingdom

REFERENCES:
- [Result] Singh D, Ciurlia G, Piccinno A, Muraro A, Bocchi M, Scuri M. Acute cardiovascular safety of two formulations of beclometasone dipropionate/formoterol fumarate in COPD patients: A single-dose, randomised, placebo-controlled crossover study. Pulm Pharmacol Ther. 2017 Feb;42:43-51. doi: 10.1016/j.pupt.2016.12.004. Epub 2017 Jan 5. PMID 28065679
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2013-002966-38
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-01535BC1-02.pdf